CLINICAL TRIAL: NCT03332381
Title: A Randomized Controlled Trial Comparing the Attention Training Technique and Mindful Self-Compassion
Brief Title: Attention Training Technique and Mindful Self-Compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/470-1
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Anxiety; Depression; Stress, Psychological
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention training technique (Active Comparator)
  Interventions: Behavioral: Attention training technique
- Mindful self-compassion (Active Comparator)
  Interventions: Behavioral: Mindful self-compassion

INTERVENTIONS:
Behavioral: Attention training technique — Attention training involves modifying metacognitive control and enhancing attention flexibility so that people can refrain from responding to intrusions with extended processing.
  Other Names: ATT
  Arms: Attention training technique
Behavioral: Mindful self-compassion — Self-compassion involves not avoiding painful or distressing feelings. Instead these experiences are held in awareness with kindness, understanding, and a sense of shared humanity.
  Other Names: MSC
  Arms: Mindful self-compassion

SUMMARY:
The design of the study is a randomized controlled trial. A total of 80 students with self-reported symptoms of stress/anxiety/depression will be invited to take part in a 3-session course consisting of either attention training or self-compassion/mindfulness based meditation. Attention training involves modifying metacognitive control and enhancing attention flexibility so that people can refrain from responding to intrusions with extended processing. Self-compassion involves not avoiding painful or distressing feelings. Instead these experiences are held in awareness with kindness, understanding, and a sense of shared humanity.

ELIGIBILITY:
Inclusion Criteria:

* self reported symptoms of stress/anxiety/depression

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of depression as assessed with the Patient Health Questionnaire-9 | Baseline, immediately after last session, 6 months after intervention
  Assesses symptoms of depression. Total score range from 0 (no depression) to 27 (very depressed). Lower values represent better outcome. Subscale scores are not used.
Change in symptoms of anxiety as assessed with the Generalized Anxiety Disorder-7 scale | Baseline, immediately after last session, 6 months after intervention
  Assesses symptoms of anxiety. Total score range from 0 (no depression) to 21 (very depressed). Lower values represent better outcome. Subscale scores are not used.

SECONDARY OUTCOMES:
Changes in self-compassion as assessed by the Self-Compassion Scale Short Form | Baseline, immediately after last session, 6 months after intervention
  Assessment of self-compassion. Total score range from 12 (no self-compassion) to 60 (high on self-compassion). Higher values represent better outcome. Subscale scores are not used.
Changes in the attention flexibility subscale of the Detached Mindfulness Questionnaire | Baseline, immediately after last session, 6 months after intervention
  Assessment of attention flexibility. Total score for attention flexibility range from 5 (no flexibility) to 25 (very flexible). Higher values represent better outcome. No other subscales are used.
Changes in mindfulness as assessed with The Five Facet Mindfulness Questionnaire | Baseline, immediately after last session, 6 months after intervention
  Assessment of mindfulness. Total score range from 20 (not mindful at all) to 100(very mindful). Higher values represent better outcome. Subscale scores are not analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Magne Flaten, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Psykologisk Institutt, Dragvoll, Trondheim, Norway